CLINICAL TRIAL: NCT07032129
Title: Sequential CAR-T Cells Targeting BCMA/GPRC5D in Patients With Relapsed/ Refractory Multiple Myeloma
Acronym: BAH2573
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Essen Biotech (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESBI202571
Record Dates: First submitted 2025-06-05; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Multiple Myeloma; Multiple Myeloma in Relapse; Multiple Myeloma Progression; Multiple Myeloma, Refractory
Keywords: Multiple myeloma; myeloma; Autoimmune Diseases; CAR-T; GPRC5D
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Autoimmune Diseases

STUDY DESIGN:
Intervention Model Description: Patients enrolled in this clinical trial will receive a carefully designed treatment regimen. Before the infusion of BCMA and GPRC5D CAR-T cells, participants will undergo preconditioning chemotherapy. This chemotherapy serves to create an optimal environment for CAR-T cell therapy to effectively target and eliminate B cells. Following chemotherapy, participants will receive the infusion of GPRC5D and BCMA CAR-T cells.
Masking Description: Open-label clinical trials are a category of clinical research where the masking is minimal or nonexistent. In such trials, both the participants and the researchers are fully aware of the treatment assignments, which means participants know the treatment they are receiving, and researchers are aware of each participant's treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19/GPRC5D CAR T cells, chemotherapy (Experimental): Patients will be administered fludarabine phosphate intravenously (IV) over a 30-minute period on days -4 to -2. Additionally, cyclophosphamide will be administered intravenously (IV) over 60 minutes on day -2. Subsequently, patients will receive BCMA/GPRC5D CAR T cells intravenously (IV) over a duration of 10-20 minutes on day 0. Patients who exhibit positive responses to the initial dose of BCMA/GPRC5D CAR T cells, do not experience unacceptable side effects, and have a sufficient quantity of cells available may be eligible to receive 2 or 3 additional doses of BCMA/GPRC5D CAR T cells.
  Interventions: Biological: BCMA/GPRC5D CAR-T cells

INTERVENTIONS:
Biological: BCMA/GPRC5D CAR-T cells — The intervention in this clinical trial involves a novel approach using BCMA/GPRC5D Chimeric Antigen Receptor T (CAR T) cells combined with chemotherapy. The goal is to assess safety and efficacy in patients with specific hematologic malignancies.
  Treatment Regimen:
  Patients in the trial will undergo the following regimen:
  Fludarabine Phosphate (Days -4 to -2): IV administration of fludarabine phosphate over 30 minutes on days -4 to -2. It's part of the preparatory regimen to enhance the body's response to CAR T-cell therapy.
  Cyclophosphamide (Day -2): IV cyclophosphamide over 60 minutes on day -2.
  BCMA/GPRC5D Chimeric Antigen Receptor T Cells (Day 0): IV administration of investigational therapy, BCMA/GPRC5D CAR T cells, over 10-20 minutes on day 0.
  Additional Doses: Eligible patients responding well to the initial BCMA/GPRC5D CAR-T cell infusion without unacceptable side effects and sufficient CAR-T cell availability may receive 2 or 3 additional doses.

SUMMARY:
This is an open, single-arm, clinical study to evaluate the efficacy and safety of chimeric antigen receptor T cell immunotherapy (CAR-T) targeting BCMA or GPRC5D or both sequentially in the treatment of Relapsed/ Refractory Multiple myeloma

DETAILED DESCRIPTION:
Chimeric antigen receptor (CAR)-modified T cells targeted against CD19 have demonstrated unprecedented successes in treating patients with hematopoietic and lymphoid malignancies. Besides CD19, many other molecules such as CD22, CD30,BCMA,CD123, etc. may have the potential to develop the corresponding CAR-T cells to treat patients whose tumors express those markers. In this study, investigators will evaluate the safety and efficacy of CAR-T targeting CD19/BCMA in patients with Autoimmune Disease. The primary goal is safety assessment including cytokine storm response and any other adverse effects. In addition, disease status after treatment will also be evaluated.

The purpose of this clinical trial is to assess the feasibility, safety, and efficacy of multiple CAR T-cell therapy that combines CAR T cells against Autoimmune Disease B Cells with CAR T cells targeting BCMA or GPRC5D or both in patients with relapsed and refractory Multiple Myeloma. The study also aims to learn more about the function of CAR T cells and their persistence in Multiple myeloma patients.

ELIGIBILITY:
Inclusion Criteria:

* Expected survival time ≥3 months;
* Subjects with recurrent/refractory Multiple Myeloma who have failed standard treatment or lack effective treatment, Including but not limited to systemic lupus erythematosus, idiopathic inflammatory myopathy, systemic sclerosis, IGG4-associated diseases, primary Sjogren's syndrome, rheumatoid arthritis, connective tissue disease-associated interstitial lung disease, immune thrombocytopenia, primary biliary cholangitis, etc.
* Histological evidence of non-suppurative destructive cholangitis and small bile duct destruction.
* Liver and kidney function, cardiopulmonary function meet the following requirements:
* Creatinine ≤1.5×ULN; (2) Electrocardiogram showed no clinically significant abnormal bands;
* Blood oxygen saturation >91% in non-oxygen state;
* Total bilirubin ≤2×ULN; ALT and AST≤2.5 x ULN; ALT and AST abnormalities due to disease, such as liver infiltration or bile duct obstruction, were determined to be less than 5×ULN. If Gilbert syndrome is diagnosed, the total bilirubin index can be relaxed to ≤3.0×ULN and the direct bilirubin ≤1.5×ULN.
* No serious mental disorders;
* Can understand this test and has signed the informed consent.

Exclusion Criteria:

* Malignant tumors other than R/R AID disease in the 5 years prior to screening, except for adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical surgery, and breast ductal carcinoma in situ after radical surgery;
* Hepatitis B surface antigen (HBsAg) positive; Hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer detection is not within the normal reference value range; Hepatitis C virus (HCV) Antibody positive and peripheral blood hepatitis C virus (HCV) RNA positive; Human immunodeficiency virus (HIV) Antibody positive; Syphilis positive;
* Serious heart disease, including but not limited to unstable angina, myocardial infarction or bypass or stent surgery (within 6 months prior to screening), congestive heart failure (NYHA classification ≥III), and severe arrhythmia;
* Systemic diseases that are deemed unstable by researchers: including but not limited to severe liver, kidney, or metabolic diseases that require drug treatment;
* Active or uncontrollable infections (except mild genitourinary and upper respiratory tract infections) that require systemic treatment within 7 days prior to administration;
* Pregnant or lactating women, and female subjects who plan pregnancy within 2 years after cell transfusion or male subjects whose partners plan pregnancy within 2 years after cell transfusion;
* Patients who received CAR-T therapy or other gene-modified cell therapy before screening;
* Participated in other clinical studies 1 month before screening;
* Evidence of central nervous system invasion during subject screening;
* Mental patients with depression or suicidal thoughts;
* Situations considered unsuitable for inclusion by other researchers.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2027-12-10 (Estimated); Study Completion 2028-12-28 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of dose-limiting toxicities (DLTs) following chemotherapy preparative regimen and infusion of CD19/BCMA chimeric antigen receptor (CAR) T cells | 28 days
  Will be recorded and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 at three dose levels until the maximum tolerated dose (MTD) is determined.

SECONDARY OUTCOMES:
Rate of successful manufacture and expansion of the CD19/GPRC5D chimeric antigen receptor (CAR) T cells | 60 days
  satisfy the targeted dose level and meet the required release specifications outlined in the Certificate of Analysis (COA)

CONTACTS AND LOCATIONS:
Locations (1):
- District One Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided